CLINICAL TRIAL: NCT07302854
Title: Intra-arterial Recombinant Human Tenecteplase Tissue-type Plasminogen Activator (rhTNK-tPA) Thrombolysis for Acute Medium Vessel Occlusion -- A Multicenter, Prospective, Randomized, Open-label, Blinded End-point Trial
Brief Title: Intra-arterial Recombinant Human Tenecteplase Tissue-type Plasminogen Activator (rhTNK-tPA) Thrombolysis for Acute Medium Vessel Occlusion
Acronym: MeVO-TNK Ⅱ
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiang Luo (Other)
Responsible Party: Sponsor-Investigator, Xiang Luo, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-IRB202512087
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke; Medium Vessel Occlusion
Keywords: Acute Ischemic Stroke; medium vessel occlusion; Intra-arterial thrombolysis; Tenecteplase
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients of this group will receive intra-arterial rhTNK-tPA thrombolysis plus standard medical treatment
  Interventions: Procedure: Intra-arterial Thrombolysis; Drug: Standard medical treatment
- Control group (Active Comparator): Patients of this group will receive standard medical treatment alone
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Procedure: Intra-arterial Thrombolysis — rhTNK-tPA（Tenecteplase）dose: 0.125 mg/kg, maximum dose: 12.5mg.
  Arms: Intervention group
Drug: Standard medical treatment — Standard medical treatment

SUMMARY:
Medium vessel occlusion (MeVO) accounts for 20-45% of acute ischemic stroke (AIS). Although patients with MeVO often present with relatively low NIHSS scores, up to one-third remain functionally dependent at follow-up despite receiving standard medical therapy, including intravenous thrombolysis. Recent randomized trials (DISTAL, ESCAPE-MeVO, DISCOUNT) have not demonstrated clinical benefit of endovascular treatment (EVT) for MeVO and have suggested higher risks of symptomatic intracranial hemorrhage and mortality, underscoring the need for safer and more targeted reperfusion strategies.

Intra-arterial thrombolysis (IAT) enables localized, high-concentration thrombolytic delivery with minimal mechanical manipulation, which may be advantageous for medium and distal vessels. Recombinant human TNK tissue-type plasminogen activator (rhTNK-tPA), a genetically engineered third-generation thrombolytic agent, has shown favorable pharmacologic properties and clinical safety in AIS, including in intra-arterial use following EVT. However, prospective evidence supporting its direct therapeutic role in MeVO-related AIS remains lacking.

This multicenter, prospective, open-label randomized controlled trial with blinded endpoint assessment is designed to evaluate the efficacy and safety of intra-arterial rhTNK-tPA thrombolysis in improving functional outcome in MeVO within 24 hours of symptom onset.

DETAILED DESCRIPTION:
This study is an investigator-initiated, multicenter, prospective, randomized, open-label, blinded-endpoint (PROBE) clinical trial designed to evaluate the efficacy and safety of intra-arterial rhTNK-tPA in improving 90-day functional outcomes in patients with MeVO stroke within 24 hours of symptom onset. The primary outcome is the proportion of patients achieving a modified Rankin Scale (mRS) score of 0-1 at 90 days. Eligible patients will be randomized in a 1:1 ratio to receive either intra-arterial rhTNK-tPA thrombolysis (0.125 mg/kg, Max 12.5mg) plus standard medical therapy or standard medical therapy alone. A total of 382 participants (191 per group) will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Pre-stroke mRS score 0-1
3. Baseline NIHSS ≥4 or symptoms deemed clearly disabling by treating physician (e.g., hemianopia, aphasia, or motor dysfunction)
4. Isolated medium distal vessel occlusion (i.e., an occlusion of the co-/non-dominant M2, the M3/M4 segment of the MCA, the A1/A2/A3 segment of the ACA or the P1/P2/P3 segment of the PCA) confirmed by CT angiography (CTA) or MR angiography (MRA)
5. Acute ischemic stroke within 24 hours of symptom onset, including wake-up stroke or unwitnessed stroke; The onset time of symptoms was defined as the last time of normal performance.
6. Acute ischemic stroke within 6-24 hours of onset, meeting at least one of the following imaging criteria:

   1. Evidence of a hypoperfusion-ischemic core mismatch on CT or MRI perfusion, defined as an ischemic core volume <50mL, hypoperfused tissue volume to ischemic core volume ratio ≥1.2, and mismatch volume ≥10 mL
   2. Evidence of a diffusion-hyperintensity mismatch, defined as absence of hyperintensity on fluidattenuated inversion recovery (FLAIR) imaging within ≥ 90% of the area of the diffusion weighted imaging (DWI) lesion)
7. The participant or legally authorized representative is capable of providing informed consent

Exclusion Criteria:

1. Evidence of intracranial hemorrhage
2. Any active bleeding (gastrointestinal, urinary, hemorrhagic retinopathy, etc.) or parenchymal organ surgery or biopsy within 30 days before stroke; Severe head trauma or stroke within the past 3 months
3. Persistent and uncontrolled hypertension, defined as systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg
4. Inherited or acquired hemorrhagic tendancy; deficiency of anticoagulant factors; or on oral anticoagulant with an INR> 1.7
5. Blood glucose <2.8 mmol/L (50 mg/dl) or > 22.2mmol/L (400 mg/dl), platelets count <100*109/L, or hemoglobin <70g/L
6. Severe hepatic insufficiency, chronic hemodialysis and severe renal insufficiency (or recent blood tests suggesting a glomerular filtration rate <30 ml/min or blood creatinine> 200 mmol/L (2.5 mg/dl)
7. Women who are pregnant or breastfeeding
8. Allergy to rhTNK-tPA or radiocontrast agent
9. Participation in other clinical trials
10. Expected survival time less than 6 months (e.g., due to malignancy, severe cardiopulmonary disease, etc.)
11. Other conditions deemed by the investigator to make the patient unsuitable for participation or pose significant risks (e.g., inability to understand and/or comply with study procedures and/or follow-up due to mental illness, cognitive or emotional disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Excellent outcome | 90±7 days
  Rate of modified Rankin scale (mRS) 0-1 at 90±7 days

SECONDARY OUTCOMES:
Ordinal distribution of mRS | 90±7 days
  The shift analysis of mRS at 90±7 days (mRS 5 and 6 merged)
Functional independence | 90±7 days
  Rate of mRS 0-2 at 90±7 days
Quality of life (EQ-5D-5L) | 90±7 days
  The EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) index score at 90±7 days
  The EQ-5D-5L is a standardized, preference-based measure of health-related quality of life covering five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five severity levels. The EQ-5D-5L index score typically ranges from less than 0 (health states worse than death) to 1.0 (full health), with higher scores indicating better quality of life.
Neurologic deficit (NIHSS score) changes | 36±12 hours
  The change of the National Institutes of Health Stroke Scale (NIHSS) score from baseline to 36±12 hours
  The NIHSS is a standardized clinical scale used to quantify neurologic impairment in stroke patients. The total score ranges from 0 to 42, with higher scores indicating more severe neurologic deficit. The outcome is defined as the change in NIHSS score from baseline, where a greater negative change reflects greater neurologic improvement.
Infarct core volume change from baseline | 7±1 days or discharge if earlier
  Infarct core volume change from baseline at 7±1 days or discharge if earlier

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage (sICH) | 48 hours
  Rate of sICH within 48 hours after randomization (Heidelberg Bleeding Classification)
All-caused mortality | 90±7 days
  All cause mortality at 90±7 days
Any intracranial hemorrhage | 48 hours
  Rate of any intracranial hemorrhage within 48 hours after randomization (Heidelberg Bleeding Classification)

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Luo, Principal Investigator — Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei 450001
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miao Z, Luo G, Song L, Sun D, Chen W, Yao X, Pan Y, Liu Y, Yuan G, Wen C, Wei M, Cai X, Yang Q, Zhou Z, Chang M, Nan G, Wang J, Xiang G, Zhou L, Gao W, Zhang H, Hao J, Xu C, Sun Y, Yi T, Feng G, Han H, Gao F, Ma N, Mo D, Sun X, Deng Y, Tong X, Li X, Jia B, Wang B, He Z, Yang M, Zhao X, Zhang X, Zhang L, Li S, Tong X, Jing J, Xiong Y, Liu T, Li Z, Ren Z, Wang Y, Liebeskind DS, Jovin TG, Nguyen TN, Wang Y, Liu L, Yan B, Huo X; ANGEL-TNK Investigators. Intra-arterial Tenecteplase for Acute Stroke After Successful Endovascular Therapy: The ANGEL-TNK Randomized Clinical Trial. JAMA. 2025 Aug 19;334(7):582-591. doi: 10.1001/jama.2025.10800. PMID 40616323
- [Background] Goyal M, Ospel JM, Ganesh A, Dowlatshahi D, Volders D, Mohlenbruch MA, Jumaa MA, Nimjee SM, Booth TC, Buck BH, Kennedy J, Shankar JJ, Dorn F, Zhang L, Hametner C, Nardai S, Zafar A, Diprose W, Vatanpour S, Stebner A, Bosshart S, Singh N, Sebastian I, Uchida K, Ryckborst KJ, Fahed R, Hu SX, Vollherbst DF, Zaidi SF, Lee VH, Lynch J, Rempel JL, Teal R, Trivedi A, Bode FJ, Ogungbemi A, Pham M, Orosz P, Abdalkader M, Taschner C, Tarpley J, Poli S, Singh RJ, De Leacy R, Lopez G, Sahlas D, Chen M, Burns P, Schaafsma JD, Marigold R, Reich A, Amole A, Field TS, Swartz RH, Settecase F, Lenzser G, Ortega-Gutierrez S, Asdaghi N, Lobotesis K, Siddiqui AH, Berrouschot J, Mokin M, Ebersole K, Schneider H, Yoo AJ, Mandzia J, Klostranec J, Jadun C, Patankar T, Sauvageau E, Lenthall R, Peeling L, Huynh T, Budzik R, Lee SK, Makalanda L, Levitt MR, Perry RJ, Hlaing T, Jahromi BS, Singh P, Demchuk AM, Hill MD; ESCAPE-MeVO Investigators. Endovascular Treatment of Stroke Due to Medium-Vessel Occlusion. N Engl J Med. 2025 Apr 10;392(14):1385-1395. doi: 10.1056/NEJMoa2411668. Epub 2025 Feb 5. PMID 39908448
- [Background] Psychogios M, Brehm A, Ribo M, Rizzo F, Strbian D, Raty S, Arenillas JF, Martinez-Galdamez M, Hajdu SD, Michel P, Gralla J, Piechowiak EI, Kaiser DPO, Puetz V, Van den Bergh F, De Raedt S, Bellante F, Dusart A, Hellstern V, Khanafer A, Parrilla G, Morales A, Kirschke JS, Wunderlich S, Fiehler J, Thomalla G, Lemmens R, Peluso JP, Bolognese M, von Hessling A, van Es A, Kruyt ND, Coutinho JM, Castano C, Minnerup J, van Zwam W, Dhondt E, Nolte CH, Machi P, Loehr C, Mattle HP, Buhk JH, Kaesmacher J, Dobrocky T, Papanagiotou P, Alonso A, Holtmannspoetter M, Zini A, Renieri L, Keil F, van den Wijngaard I, Kagi G, Terceno M, Wiesmann M, Amaro S, Rommers N, Balmer L, Fragata I, Katan M, Leker RR, Saver JL, Staals J, Fischer U; DISTAL Investigators. Endovascular Treatment for Stroke Due to Occlusion of Medium or Distal Vessels. N Engl J Med. 2025 Apr 10;392(14):1374-1384. doi: 10.1056/NEJMoa2408954. Epub 2025 Feb 5. PMID 39908430